CLINICAL TRIAL: NCT03506256
Title: Noroxin Efficacy and Safety Trial
Acronym: NEST
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: OBS Pakistan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBS-NEST-003
Record Dates: First submitted 2018-04-01; First posted 2018-04-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Urinary Tract Infections
Keywords: urinary tract infection; Norfloxacin; Fluroquinolone; Safety; Pakistan
MeSH Terms: conditions — Urinary Tract Infections | interventions — Norfloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Norofloxacin (Experimental): The recommended dosage of norfloxacin for urinary-tract infections in adults is 400 mg orally every 12 hours; the drug should be given for 7 to 10 days in uncomplicated infections and for 10 to 21 days in complicated ones. Adverse drug effects were mild and included disturbances of the gastrointestinal tract and the central nervous system. The study shall be completed in accordance with the ICH topic E6 (R1)(CPMP/ICH/one hundred thirty five/95) guiding principle for top medical practice and the ideas enunciated within the announcement of Helsinki and the approval by way of an Institutional Ethics Committee.
  Interventions: Drug: Norfloxacin 400 MG

INTERVENTIONS:
Drug: Norfloxacin 400 MG — Norfloxacin is an oral fluoroquinolone antimicrobial agent used for the treatment of uncomplicated and complicated urinary tract infections. The drug antagonizes DNA gyrase, an enzyme essential for bacterial DNA replication and is active in vitro against virtually all bacterial pathogens causing urinary tract8

SUMMARY:
To determine the efficacy and safety of Norfloxacin (Noroxin)

DETAILED DESCRIPTION:
Urinary tract infections (UTIs) are some of the most common bacterial infections, affecting 150 million people each year worldwide. Clinically, UTIs are categorized as uncomplicated or complicated. Uncomplicated UTIs typically affect individuals who are otherwise healthy and have no structural or neurological urinary tract abnormalities; these infections are differentiated into lower UTIs (cystitis) and upper UTIs (pyelonephritis). Several risk factors are associated with cystitis, including female gender, a prior UTI, sexual activity, vaginal infection, diabetes, obesity and genetic susceptibility.

UTIs are caused by both Gram-negative and Gram-positive bacteria, as well as by certain fungi. The most common causative agent for both uncomplicated and complicated UTIs is uropathogenic Escherichia coli (UPEC). For the agents involved in uncomplicated UTIs, UPEC is followed in prevalence by Klebsiella pneumoniae, Staphylococcus saprophyticus, Enterococcus faecalis, group B Streptococcus (GBS), Proteus mirabilis, Pseudomonas aeruginosa, Staphylococcus aureus and Candida spp. Currently, antibiotics - such as trimethoprim sulfamethoxazole, floxacin and ampicillin - are the most commonly recommended therapeutics for UTIs6. UTIs are becoming increasingly difficult to treat owing to the widespread emergence of an array of antibiotic resistance mechanisms. Of particular concern are members of the family Enterobacteriaceae, including E. coli and K. pneumoniae, which have both acquired plasmids encoding extended-spectrum β-lactamases (ESBLs). These plasmids rapidly spread resistance to third-generation cephalosporins as well as other antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* At least one typical symptom of acute, lower urinary tract infection out of dysuria, frequency, macrohaematuria, cloudy or smelly urine or self-diagnosed cystitis

Exclusion Criteria:

* Duration of UTI symptoms for more than 7 days before physician's visit
* Clinical signs of invasiveness such as fever (axillary body temperature >38 degrees Celsius), costovertebral pain or tenderness, rigors, nausea or vomiting
* Known or suspicion of anatomical or functional abnormality of the urinary tract
* Vaginal symptoms: discharge, irritation
* Diabetes mellitus
* Immunosuppression (e.g. prednisone equivalent >10mg per day for >14 days, chemotherapy, radiotherapy, immunomodulators, HIV infection, neutropenia)
* Any other serious comorbidity as judged by the treating physician
* Bladder catheter in situ or during the past 30 days
* Pregnancy
* Recurrent urinary tract infection (more than 3 infections during the last 12 months)
* Antibiotic treatment during the last 4 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-05-10 (Estimated); Primary Completion 2018-06-10 (Estimated); Study Completion 2018-07-30 (Estimated)

PRIMARY OUTCOMES:
Number of Patients treated with Noroxin (Efficacy) | 14 Days
  To evaluate efficacy of Norfloxacin by measuring clinical response, the resolution of sign and symptoms of post-therapy as compared to start of therapy

SECONDARY OUTCOMES:
Number of Adverse Effects with Noroxin (Safety) | 14 Days
  To determine number of patients that experienced Adverse effects

IPD SHARING:
Plan to Share IPD: No